CLINICAL TRIAL: NCT05184296
Title: ExtraCorporeal Membrane Oxygenation in the Therapy for REfractory Septic Shock With Cardiac Function Under Estimated (ECMO-RESCUE): a Prospective, Multicenter, Non-randomized Cohort Study
Brief Title: ExtraCorporeal Membrane Oxygenation in the Therapy for REfractory Septic Shock With Cardiac Function Under Estimated
Acronym: ECMO-RESCUE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICU-02
Record Dates: First submitted 2021-12-20; First posted 2022-01-11 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-11

CONDITIONS: Extracorporeal Membrane Oxygenation; Septic Shock; Septic Cardiomyopathy; Cardiogenic Shock
Keywords: Extracorporeal Membrane Oxygenation; refractory septic shock; septic cardiomyopathy; cardiogenic shock
MeSH Terms: conditions — Shock, Septic; Shock, Cardiogenic | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cohort 1 (Experimental): Participants taking VA-ECMO during the period of study are referred to as cohort 1
  Interventions: Procedure: Extracorporeal Membrane Oxygenation (ECMO)
- cohort 2 (No Intervention): Patients receiving only conventional therapy without ECMO belong to cohort 2

INTERVENTIONS:
Procedure: Extracorporeal Membrane Oxygenation (ECMO) — All patients in cohort 1 will initiate ECMO as fast as possible. A maximum of 6 hours is allowed between enrollment and the actual initiation of ECMO. ECMO catheterization and management will be operated by an experienced ECMO team and carried out at the bedside. VA or VAV mode will be chosen according to the patient's condition.
  Arms: cohort 1

SUMMARY:
The ECMO-RESCUE study is a prospective, multicenter, non-randomized, cohort study. In this study, we aimed to assessed whether VA-ECMO treatment can improve the 30-day survival rate of patients with sepsis-induced refractory cardiogenic shock.

DETAILED DESCRIPTION:
All patients who meet inclusion criteria and have no exclusion criteria are considered to be enrolled. During the period of study, the participants can decide whether to accept ECMO based on their personal conditions. If a patient is willing to accept ECMO treatment, we initiate VA-ECMO within 6 hours. Participants taking VA-ECMO during the period of study are referred to as cohort 1, and patients receiving only conventional therapy without ECMO belong to cohort 2. 30-day survival will be accessed to evaluate the survival benefit from ECMO therapy for sepsis-induced refractory cardiogenic shock.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years.
* Patients admitted into ICU and diagnosed as septic shock (sepsis-3.0)13, after adequate fluid resuscitation, high-dose vasoactive drug application [vasoactive inotropic score (VIS) > 120] and conventional therapy together with at least one of the following criteria: (1) sustained hypotension [mean arterial pressure (MAP) < 65 mmHg]; (2) persistent lactacemia (two consecutive values > 5 mmol/L with at least 30 min interval between samples), with non-decreasing trend on steady doses of inotropes and/or vasopressors; (3) persistent low mixed venous blood oxygen saturation (SvO2) (two consecutive values < 55% with at least 30 min interval between samples), with non-increasing trend on steady doses of inotropes and/or vasopressors. The above condition lasts more than 5 hours.
* Rapidly deteriorating sepsis-induced myocardial impairment is defined by at least one of the following criteria: (1) rapidly deteriorating ventricular function (LVEF < 35%); (2) cardiac index (CI) < 2L/min/m2 (> 3 hr); (3) emerging refractory arrhythmia.
* Informed consent provided by the patient or person with decisional responsibility.

Exclusion Criteria:

* Cardiac dysfunction caused by other causes is excluded, such as acute myocardial infarction, chronic heart failure, congenital cardiac disease, myocardial effusion, moderate to severe aortic regurgitation, severe aortic coarctation and so on.
* High suspicion of pulmonary embolism, tension pneumothorax or cardiac tamponade as a cause of shock.
* Prolonged cardiac arrest (> 30 min) before ECMO, or CPR survivors remaining comatose.
* Irreversible condition or meet the inclusion criteria for more than 12 hr.
* Presence of active bleeding or anticoagulant contraindications.
* Peripheral artery disease disabling insertion of outflow cannula to femoral artery.
* Irreversible neurological pathology
* Severe underlying condition with lift expectancy less than 1 year.
* Special population, such as pregnancy, acquired immune deficiency syndrome (AIDS).
* Patient included in another interventional clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
30-day survival | From date of enrolled (D0) until date of death from any cause or day-30, whichever came first
  survival rate at day-30

SECONDARY OUTCOMES:
ICU survival rate | From date of enrolled (D0) until date of death from any cause or date of discharge from ICU, whichever came first, assessed up to 6 months
  survival to ICU discharge
hospital survival | From date of enrolled (D0) until date of death from any cause or date of discharge from hospital, whichever came first, assessed up to 6 months
  survival to hospital discharge
6-month survival | From date of enrolled (D0) until the date of death from any cause or 6-month, whichever came first
  survival rate at 6-month
quality of life for long-term survival | at 6-months
  evaluate through EuroQol Five Dimensions Questionnaire Descriptive System at 6-month within survivors, the minimum value is 3, the maximum value is 15, higher scores mean a worse state.
successful rate of ECMO weaning | From date of weaning off ECMO until the date of death or 24 hours after ECMO weaning, whichever came first
  Successful weaning is defined as maintaining stable condition within 24 hours of ECMO weaning. Analyzed the frequency of patients who weaning ECMO successfully
long-term survivors' cardiac function | at day-30 and 6-month
  LVEF evaluated according to Doppler echocardiography
the number of days alive without CRRT, mechanical ventilation and vasopressor | between Day 0 and up to Day 30
  the numbers of CRRT-free days, mechanical ventilation-free days and vasopressor-free days
ICU length of stay (LOS) | From date of enrolled (D0) until the date of death from any cause or discharge from ICU, whichever came first, assessed up to 6 month
  ICU LOS
hospital length of stay (LOS) | From date of enrolled (D0) until the date of death from any cause or discharge from hospital, whichever came first, assessed up to 6 month
  hospital LOS

OTHER OUTCOMES:
safety assessments | from the date of enrolled (D0) until death or day-30, whichever came first.
  the rate of complications potentially related to ECMO treatment, including major bleeding associated with anticoagulants, thrombosis, leg ischemia and cannulation-related injuries.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen-hui Zhang, Study Director — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Chen Weiyan, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen WY, Guo ZB, Kong TY, Chen WX, Chen XH, Yang Q, Wen YC, Wen QR, Zhou F, Xiong XM, Wen DL, Zhang ZH. ExtraCorporeal Membrane Oxygenation in the therapy for REfractory Septic shock with Cardiac function Under Estimated (ECMO-RESCUE): study protocol for a prospective, multicentre, non-randomised cohort study. BMJ Open. 2024 Jun 10;14(6):e079212. doi: 10.1136/bmjopen-2023-079212. PMID 38858161